CLINICAL TRIAL: NCT00055094
Title: Immune Control of HIV Replication
Brief Title: Treatment of Acute HIV Infection to Preserve Immune Function
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 1R01AI044656-01 (NIH); 5R01AI044656-04 (NIH)
Record Dates: First submitted 2003-02-19; First posted 2003-02-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: HIV Infections
Keywords: Immune system; Helper T-Cells; Acute Infection; Treatment naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
While most people with HIV experience significant destruction of their immune systems, some people appear to have preserved immune function and can control the virus without drugs. Early treatment with anti-HIV drugs may help preserve the immune system, allowing it to control the virus once the drugs are stopped. This study will evaluate the immune system response of HIV infected people who are treated with anti-HIV drugs soon after being infected.

DETAILED DESCRIPTION:
Studies have identified a potent CD4 T helper (Th) cell response in some infected people, and have shown a correlation between virus-specific Th cells and low levels of viremia. Early institution of potent antiviral therapy in the earliest stages of acute HIV infection have led to strong Th cell responses, analogous to those seen in people who are able to control viremia in the absence of antiviral therapy. This may be because potent antiviral therapy is able to protect virus-specific Th cells as they become activated, and thus these cells are not lost in the earliest stages of infection. This study will characterize the immune response of patients with acute HIV infection who receive antiretroviral therapy and will determine the effects of interruption of therapy in those people who have immune responses to HIV that are similar to patients with long-term non-progressing infection.

Participants in this study will be followed through June 2004. Study visits vary from only once to every month and are scheduled at the discretion of the study officials. Study visits include an interview and blood tests.

ELIGIBILITY:
Inclusion Criteria

* Acute HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Walker, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States